CLINICAL TRIAL: NCT04153578
Title: Time to Lose the Weight? Comparison of Weight-based and Non-weight-based Vasopressors for Septic Shock
Status: Completed | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 057.PHA.2019.A
Record Dates: First submitted 2019-11-04; First posted 2019-11-06 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Septic Shock; Weight, Body
MeSH Terms: conditions — Shock, Septic; Body Weight

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
At present, there is conflicting evidence regarding outcomes in patients with septic shock receiving weight-based vasopressor (WBVP) versus non-weight-based vasopressor (NWBVP) dosing strategies. At MCMC, a weight-based strategy is in place whereas MDMC, MMMC and MRMC currently utilize a non-weight-based dosing strategy. Obese patients (BMI > 30) receiving either strategy may potentially be receiving substantially more or less vasopressor exposure compared to their non-obese (BMI < 30) counterparts. Determining total vasopressor exposure and assessing clinical outcomes would benefit our institution and others by providing optimal vasopressor dosing strategies in obese and non-obese patients. There is a difference in clinical outcomes between patients receiving weight-based and non-weight-based vasopressor dosing strategies. There is a difference in total vasopressor exposure between obese and non-obese patients utilizing WBVP and NWBVP strategies.

DETAILED DESCRIPTION:
Vasopressors are a mainstay of therapy for patients with septic shock to achieve and maintain hemodynamic stability.1 Both weight-based and non-weight-based dosing recommendations exist with no clear evidence that one is better than the other.3-10 However, in light of the obesity epidemic and emerging evidence regarding the dangers of excessive catecholamine exposure, an evaluation of dosing practices is warranted. The aim of this study is to determine whether clinical outcomes differ between patients receiving weight-based and non-weight-based vasopressor dosing strategies for septic shock. This is a multicenter, retrospective chart review. Patients admitted to MDMC and MCMC from 4/1/2017-8/31/2019 will be identified through the electronic medical record utilizing ICD codes for sepsis and septic shock. Patients meeting study inclusion criteria will be analyzed as described below. Outcomes will be assessed between patients receiving WBVP and NWBVP with planned subgroup analysis in each group between patients with BMI < 30, 30-49, and > 50.

ELIGIBILITY:
Inclusion Criteria:

* ICU admission
* Medical admission type
* Received NE, epinephrine (EPI), phenylephrine (PE), or dopamine (DA) for septic shock
* Received NE/EPI/PE/DA for > 24 hours
* Age ≥ 18 years

Exclusion Criteria:

* Non-sepsis indication for vasopressors
* Surgical or trauma admission type
* ICU length of stay < 24 hours
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to MDMC and MCMC from 4/1/2017-8/31/2019 will be identified through the electronic medical record utilizing ICD codes for sepsis and septic shock.
Sampling Method: Non-Probability Sample
Enrollment: 945 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2020-06-22 (Actual); Study Completion 2020-06-22 (Actual)

PRIMARY OUTCOMES:
Efficacy: Total 48-hour vasopressor exposure | 4/1/2017-8/31/2019
  Total 48-hour vasopressor exposure (norepinephrine (NE) equivalents, mg)
Safety: Composite of in-hospital mortality, vasopressor-associated adverse events | 4/1/2017-8/31/2019
  Composite of in-hospital mortality, vasopressor-associated adverse events (arrhythmia, thrombosis)

SECONDARY OUTCOMES:
Efficacy: Total number of vasoactive agents required to maintain mean arterial pressure | 4/1/2017-8/31/2019
  Total number of vasoactive agents required to maintain mean arterial pressure (MAP) > 65 mmHg, time to hemodynamic stability, use of angiotensin II or vasopressin
Safety: in-hospital mortality, vasopressor-associated adverse events | 4/1/2017-8/31/2019
  in-hospital mortality, vasopressor-associated adverse events (arrhythmia, thrombosis)

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Reiter, PharmD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided